CLINICAL TRIAL: NCT01507766
Title: The Correlations Between Early Enteral Nutrition and Intra-abdominal Pressure in Severe Acute Pancreatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Collaborators: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jiakui Sun, Principal Investigator, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 110-85
Record Dates: First submitted 2012-01-03; First posted 2012-01-11 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Acute Pancreatitis; Intra-abdominal Hypertension
Keywords: severe acute pancreatitis; intra-abdominal pressure; enteral nutrition
MeSH Terms: conditions — Pancreatitis; Intra-Abdominal Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early enteral nutrition (Experimental): The enteral nutrition was started within 48h after admission
  Interventions: Drug: early enteral nutrition
- Delayed enteral nutrition (Active Comparator): The enteral nutrition was started at the 8th day after admission
  Interventions: Drug: Delayed enteral nutrition

INTERVENTIONS:
Drug: early enteral nutrition — The enteral nutrition was started within 48h after admission
  Arms: Early enteral nutrition
Drug: Delayed enteral nutrition — The enteral nutrition was started at the 8th day after admission
  Arms: Delayed enteral nutrition

SUMMARY:
As an important management of severe acute pancreatitis (SAP), enteral nutrition (EN), especially early enteral nutrition (EEN) increases the blood flow of gut mucosa and stimulates the intestinal motility. Moreover, EEN maintains the gut integrity, prevents bacterial and endotoxin translocation and thereby theoretically reduces the incidence of infections. Therefore, EEN has the ability to reduce the infectious complications, length of hospital stay and mortality of patients with SAP.

However, the role of EEN is considered to be influenced by intra-abdominal hypertension (IAH) in patients with SAP. The previous studies showed that gut was the most sensitive splanchnic organ to the increase of intra-abdominal pressure (IAP). When IAH occurs, it reduces the blood flow of gut, and then results in the development of intestinal ischemia and edema. The hypoxia and hypoperfusion of intestine leads to the increase of permeability of the intestinal mucosal barrier, and then leads to bacterial translocation. Therefore, IAH could result in the gastrointestinal dysfunction. Nevertheless, the different impacts of specific IAP values on the tolerance of EEN have not been reported.

Furthermore, the effects of early enteral feeding on the IAP in SAP also remain unknown. Due to the severe inflammatory response of SAP, could EEN increase the burden of bowel, cause expansion of intestinal cavity, thus increase IAP? However, there were rare literatures up to date reporting the association between EEN and IAH in patients with SAP. Therefore, the present study aimed to investigate the influence of specific IAP on the tolerance of early enteral feeding, as well as the effects of EEN on IAP in SAP patients. Moreover, the impacts of EEN on the disease severity and clinical outcome of SAP were also researched.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of acute pancreatitis accords with the Atlanta criteria in 1992
* Within 3 days from the onset of the disease
* Hemodynamics stable

Exclusion Criteria:

* Decompressive measures and enteral nutrition was performed before admission
* Ileus of lower digestive tract
* Pregnant pancreatitis
* Chronic organs dysfunction
* Immunodeficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Enteral nutrition | 14 days
  The caloric intake and tolerance of feeding were recorded daily after enteral nutrition was started
Intra-abdominal pressure | 14 days
  The value of intra-abdominal pressure (per 6 hours) and the incidence of intra-abdominal hypertension

SECONDARY OUTCOMES:
Clinical outcome variables | 14 days
  Hospital mortality; Duration of ICU stay; The development of multiple organ dysfunction syndrome and pancreatic infection; APACHEII score; SOFA score; CRP levels
Immune parameters | 14 days
  IgA, IgG, IgM, CD4+/CD8+T cell and HLA-DR

CONTACTS AND LOCATIONS:
Overall Officials: Wei-qin Li, M.D., Study Director — Jinlin Hospital
Locations (1):
- Department of SICU, Research Institute of General Surgery , Jinling Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Sun JK, Li WQ, Ke L, Tong ZH, Ni HB, Li G, Zhang LY, Nie Y, Wang XY, Ye XH, Li N, Li JS. Early enteral nutrition prevents intra-abdominal hypertension and reduces the severity of severe acute pancreatitis compared with delayed enteral nutrition: a prospective pilot study. World J Surg. 2013 Sep;37(9):2053-60. doi: 10.1007/s00268-013-2087-5. PMID 23674254
- [Derived] Sun JK, Mu XW, Li WQ, Tong ZH, Li J, Zheng SY. Effects of early enteral nutrition on immune function of severe acute pancreatitis patients. World J Gastroenterol. 2013 Feb 14;19(6):917-22. doi: 10.3748/wjg.v19.i6.917. PMID 23431120